CLINICAL TRIAL: NCT07032974
Title: Prospective Randomized Controlled Trial Comparing Accuracy Among Franseen, Forward-bevel Westcott, and Fork-tip Needle Design for EUS-guided Fine Needle Biopsy in Diagnosis of Solid Pancreatic Lesions
Brief Title: RCT Comparing Accuracy Among Franseen, Forward-bevel Westcott, and Fork-tip EUS-FNB Needle in Diagnosis of Solid Pancreatic Lesions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Varayu Prachayakul, Associate Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: Si 316/2022
Record Dates: First submitted 2025-06-12; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Masses
Keywords: Pancreatic mass; EUS; EUS-FNB; Fine needle biopsy; Endoscopic ultrasound; Pancreatic lesion

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes

ARMS (3):
- Franseen (Experimental)
  Interventions: Device: Franseen
- Forward- bevel (Experimental)
  Interventions: Device: Forward-bevel
- Fork-tip (Experimental)
  Interventions: Device: Fork-tip

INTERVENTIONS:
Device: Franseen — Franseen needle
  Arms: Franseen
Device: Forward-bevel — Forward-bevel needle
  Arms: Forward- bevel
Device: Fork-tip — Fork-tip needle
  Arms: Fork-tip

SUMMARY:
Endoscopic Ultrasound-Guided Fine Needle Aspiration (EUS-FNA) is a well-established technique for pancreatic tissue acquisition, offering a high diagnostic accuracy ranging from 78% to 95%, along with a favorable safety profile. Over time, numerous studies have sought to optimize this procedure by investigating various contributing factors, including needle size, sampling techniques, adequacy of tissue acquisition, the number of passes required, and needle type. These insights have largely been incorporated into routine clinical practice, refining the diagnostic capabilities of EUS-FNA.

Despite its widespread use, EUS-FNA has limitations, particularly in the diagnosis of certain pancreatic pathologies such as lymphoma, gastrointestinal stromal tumors (GISTs), and autoimmune pancreatitis. These conditions often require histologic samples for ancillary studies, which cytologic specimens obtained via FNA cannot sufficiently provide. To overcome this limitation, Fine Needle Biopsy (FNB) needles were developed. These needles enable the procurement of core tissue samples, thereby enhancing histopathological assessment and reducing reliance on rapid on-site cytological evaluation (ROSE). Additionally, FNB allows for fewer needle passes, which can shorten procedure time and reduce associated complications.

Among FNB technologies, the third generation of needles has garnered particular attention due to improved sample adequacy and diagnostic reliability. While earlier research compared second-generation FNB needles with FNA, demonstrating no significant difference in diagnostic yield, more recent studies suggest that third-generation FNB needles offer superior diagnostic accuracy.

Currently, three distinct third-generation FNB needle types are commercially available, distinguished by their tip geometry:

Franseen geometry - Acquire™ (Boston Scientific)

Fork-tip - SharkCore™ (Medtronic)

Forward-bevel Westcott - ProCore™ (Cook Medical)

Despite their clinical adoption, comparative data on their diagnostic performance remain scarce. Only two randomized controlled trials (RCTs) have directly compared these needle types:

Karsenti et al. compared the Franseen (Acquire) and the Forward-bevel Westcott (ProCore) needles for pancreatic mass diagnosis. Diagnostic accuracy was 87% (CI: 75-94) for the Franseen needle and 67% (CI: 53-78) for the Westcott needle, with a statistically significant difference (p = 0.02).

Ashat et al. evaluated the Franseen (Acquire) and Fork-tip (SharkCore) needles in diagnosing all gastrointestinal masses, reporting diagnostic accuracies of 85.3% and 90.7%, respectively (p = 0.45). In a pancreatic mass-specific subgroup analysis, accuracy rates were 89.7% and 94.4%, respectively (p = 0.68), suggesting comparable performance between the two.

Despite these findings, the current literature does not include a comprehensive head-to-head comparison encompassing all three third-generation FNB needle types. Therefore, it remains uncertain which design offers the best diagnostic performance for pancreatic tumors. The absence of such comparative studies presents a significant gap in the field of EUS-guided tissue acquisition.

DETAILED DESCRIPTION:
Endoscopic Ultrasound-Guided Fine Needle Aspiration (EUS-FNA) for pancreatic tissue acquisition is a widely accepted and popularly used technique because of its high diagnostic accuracy of 78% - 95% and a low risk of adverse events.

Previous studies have tried to identify ways to increase the efficacy and diagnostic accuracy of EUS-FNA. Many factors were found to influence the diagnostic accuracy of EUS-FNA which included needle size, sampling technique, evaluation of tissue adequacy, number of needle passes, and finally the needle type, which the impact of most of the aforementioned factors were thoroughly studied and already incorporated into the standard practice of pancreatic tissue acquisition.

It was difficult to diagnose some pancreatic diseases by EUS-FNA, such as lymphoma, gastrointestinal stromal tumor (GIST), and autoimmune pancreatitis because the cytologic specimen was simply not enough for further ancillary studies. FNB needles were subsequently developed to eliminate this limitation, by obtaining a larger specimen, FNB needles enable pathologists to evaluate the specimens more thoroughly and help guide further therapeutic decisions. In addition, it reduces the dependency on immediate cytological examination during endoscopy (Rapid on-site evaluation [ROSE]) and also reduces the procedure duration, since the number of needle passes is reduced.

The continuous development of EUS-FNB needles has been a major area of interest in recent years. In particular, the third generation of FNB needles were developed to obtain a more adequate tissue sample. Previous research has focused on comparing the accuracy of the second generation FNB needles with the FNA needles in the diagnosis of pancreatic tissue. Results from these studies found no significant differences between the two needles. However, it was discovered that the third generation FNB needle has significantly higher diagnostic accuracy than the FNA needle. These findings suggest that the third generation FNB needle may be a more reliable and effective tool for diagnosing tissue samples in various clinical settings.

In the field of tissue biopsy, the third generation FNB needle is currently available in three types based on the characteristics of the needle tip. These types include Franseen geometry needle (Acquire, Boston Scientific), Fork-tip needle (Shark-core, Medtronic), and Forward-bevel Westcott (Procore, Cook Medical). However, there is a lack of research comparing the diagnostic accuracy of among each type of needle. Only two randomized controlled trials have been conducted to address this issue. Karsenti et al. investigated the accuracy of diagnosing a pancreatic mass using Franseen geometry needle (Acquire, Boston Scientific) and Forward-bevel Westcott (Procore, Cook Medical). The study found accuracy rates of 87% (75-94) and 67% (53-78), respectively, with a p-value of 0.02. Ashat et al. compared the accuracy of diagnosing all gastrointestinal masses using Franseen geometry needle (Acquire, Boston Scientific) and Fork-tip needle (Shark-core, Medtronic), finding accuracy rates of 85.3% and 90.7%, respectively, with a p-value of 0.45. Subgroup analysis for pancreatic masses alone found accuracy rates of 89.7% and 94.4%, respectively, with a p-value of 0.68.

In the context of diagnosing pancreatic tissue masses, only a limited number of studies have examined the comparative accuracy of 3rd generation fine needle biopsy (FNB) needles. As such, it remains unclear which type of needle can deliver superior diagnostic precision, and to date, no study has conducted a head-to-head comparison of all three needle types. Thus, the purpose of the present investigation is to assess the diagnostic accuracy of all three 3rd generation FNB needle types in the context of detecting pancreatic tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Solid pancreatic mass greater than 1 cm in size who required tissue diagnosis

Exclusion Criteria:

* Pregnancy
* Uncorrected coagulopathy
* Surgically altered anatomy
* Unable to complete informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | 6 months
  Diagnostic accuracy of three third-generation fine-needle biopsy (FNB) needles

SECONDARY OUTCOMES:
Number of needle passes | During procedure
  Number of needle passes during EUS
Overall satisfaction | During procedure
  Overall satisfaction of endoscopist during EUS including needle visiblity, maneuverability and ease of puncture on a scale of 0 to 2.
Procedure time | During procedure
  Procedure time of EUS
Adverse events | up to 2 weeks
  Adverse events of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Varayu Prachayakul, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
We are willing to provide our data to researchers who require it. For example, those who want to do systematic review and meta-analysis.
Supporting Information: Study Protocol
Time Frame: Other researchers can contact us anytime.
Access Criteria: We will provide our protocol and/or data upon request.